CLINICAL TRIAL: NCT00919451
Title: A Pilot Study Assessing the Efficacy and Safety of Ciclosporin as a Second -Line Drug in Patients With Type 1 Reactions Who Have Not Responded to a 12 Week Course of Prednisolone.
Brief Title: Ciclosporin in the Management of Steroid Resistant Type 1 Reactions in Leprosy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Homes and Hospitals of St Giles (Other); Alert Hospital, Ethiopia (Other); Armauer Hansen Research Institute, Ethiopia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITCRBY24-T1RB
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2014-09

CONDITIONS: Leprosy
Keywords: Leprosy; Type 1 Reaction; Prednisolone; Ciclosporin
MeSH Terms: conditions — Leprosy | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ciclosporin (Experimental): ciclosporin reducing regimen lasting 24 weeks (additional prednisolone given for the first four weeks)
  Interventions: Drug: ciclosporin

INTERVENTIONS:
Drug: ciclosporin — Ciclosporin 7.5mg/kg - reducing regimen over 24 weeks (additional prednisolone given for the first four weeks)

SUMMARY:
Study 1B: Ciclosporin in the management of steroid resistant Type 1 Reactions in Leprosy

Objective: A pilot study assessing the efficacy and safety of Ciclosporin as a second -line drug in patients with Type 1 Reactions who have not responded to a 12 week course of Prednisolone.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with clinical evidence of Type 1 Reaction who have not responded to 3 months Prednisolone Treatment
* Aged 18-65
* Weigh more than 30Kg

Exclusion Criteria:

* Unwillingness to give informed consent
* Patients with severe active infections such as tuberculosis
* Pregnant or breastfeeding women (see Appendix II)
* Those with renal failure, abnormal renal function, hypertensive
* Patients taking thalidomide currently or within the last 3 months
* Patients not willing to return for follow-up
* Women of reproductive age not willing to use contraception for the duration of the study ( see Appendix II)
* HIV positive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
improvement in nerve function | at 24 weeks and 32 weeks

SECONDARY OUTCOMES:
incidence of adverse effects | throughout 32 weeks
Skin lesion inflammation improvement | up to 36 weeks
rate of improvement of reaction | up to 36 weeks
Time to next reactional episode | up to 2 years
extra prednisolone needed to control reaction | up to 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diana NJ Lockwood, MBChB, Principal Investigator — London SHTM
Locations (1):
- Alert Hospital, Addis Ababa, Ethiopia